CLINICAL TRIAL: NCT05494372
Title: Assessment of Intraoperative Nursing Safety Precautions for Open Heart Surgery Patients on Cardiopulmonary Bypass Machine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Taha Badwy, Head of nurse, Assiut University
Other Study IDs: Nursing safety on CBP
Record Dates: First submitted 2022-08-05; First posted 2022-08-10 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Nursing Safety on Cardiopulmonary Bypass
Keywords: nursing safety precautions; cardiac surgery; cardiopulmonary bypass machine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Other: safety precautions — Nursing safety precautions on CPB

SUMMARY:
Assessment of intraoperative nursing safety precautions for open heart surgery patients on cardiopulmonary bypass machine.

DETAILED DESCRIPTION:
Coronary artery bypass grafts surgery (CABG) can be performed either with cardiopulmonary bypass (CPB), which exposes the blood to a non-physiological environment, or on beating heart without CPB support. One of the most challenging aspects of coronary artery bypass grafting surgery is the management of high-risk patients and management of possible complications due to cardiopulmonary bypass machine to achieve acceptable morbidity, mortality, and quality of life Nursing safety precautions during cardiopulmonary bypass surgery begins with the perfusionists and critical care nurses experience and knowledge of all the possible errors that may occur. This knowledge fosters the anticipation of problems and promotes vigilance safety precautions for prevention of possible complications which may occur as a result of cardiopulmonary bypass machine.

Advances in cardiac surgery have been possible due to the development of cardiopulmonary bypass machine. Cardiopulmonary bypass machine is a form of extracorporeal circulation whose function is circulatory and respiratory support along with temperature management to facilitate surgery on the heart and great vessels. The first successful human cardiac surgery using CPB was performed by John Gibbon in 1952 for repair of the atrial septal defect. Complications that occur as a result of cardiopulmonary bypass machine in cardiac surgery patients includes mechanical and systemic complications, mechanical complications such as bleeding, oxygenator failure, pump malfunction, clotting in the circuit, tubing rupture, gas supply failure and electrical failure. Systemic complications include qualitative and quantitative platelet dysfunction. Inflammatory response and hypotension can cause acute kidney injury. Risk factors are prolonged bypass time, sepsis and diabetes. cerebral injury ranges from cognitive dysfunction to stroke. Acute respiratory distress syndrome can be present due to the effects of CPB.

Nursing safety precautions related to cardiac surgery with cardiopulmonary bypass machine were written with collaboration from the Society of Cardiovascular Anesthesiologists, and an update to these safety precautions that have collaborated on nursing safety precautions for anticoagulation, as Clotting on cardiopulmonary bypass is life-threatening. Temperature management, acid base balance management, monitoring on cardiopulmonary bypass, ultra-filtration during and after CPB removes inflammatory mediators and weaning management. These safety precautions provide professional nurses with actionable evidence informed by expert opinion, to achieve acceptable morbidity, mortality, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60years.
* Coronary artery bypass grafting patients.
* Aortic valve replacement/repair patients.
* Mitral valve replacement/repair patients.
* Tricuspid valve replacement/repair patients.
* In addition to critical care nurses whom are also willing to participate in this study.

Exclusion Criteria:

The exclusion criteria are as follow:

* patients with previous open-heart surgery.
* Patients with high bleeding tendency.
* patients with associated aneurysm of the left ventricle or ischemic VSD defect with recent cardiac infarction.
* patients with liver cell failure.
* Patients with renal failure on regular dialysis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Convenient sample of 60 adult male and female patients who presented to cardiothoracic unit for undergoing cardiac surgery using cardiopulmonary bypass machine were included in addition to 20 critical care nurses acts as a perfusionist who are willing to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-09-04 (Actual); Primary Completion 2022-09-10 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
assessment of nursing safety precautions for cardiac surgery patients on cardiopulmonary bypass machine | baseline
  * This part was including assessment of nursing safety precautions during surgery for patients on cardiopulmonary bypass machine using scoring system.
  * Nursing safety precautions consists of four main items each item divided into steps, each step takes a score ranging from 0 to 2, minimum score is 0 (not apply), medium score is1 (need improve) and maximum score is 2 (well done).
  * Total steps in four items are 45 steps their total score is 90, scoring system transformed into percent:( < 85% unsatisfactory), (>= 85% satisfactory).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Asyut, Egypt

REFERENCES:
- [Background] Rijkse E, de Jonge J, Kimenai HJAN, Hoogduijn MJ, de Bruin RWF, van den Hoogen MWF, IJzermans JNM, Minnee RC. Safety and feasibility of 2 h of normothermic machine perfusion of donor kidneys in the Eurotransplant Senior Program. BJS Open. 2021 Jan 8;5(1):zraa024. doi: 10.1093/bjsopen/zraa024. PMID 33609374
- [Background] Jochmans I, Brat A, Davies L, Hofker HS, van de Leemkolk FEM, Leuvenink HGD, Knight SR, Pirenne J, Ploeg RJ; COMPARE Trial Collaboration and Consortium for Organ Preservation in Europe (COPE). Oxygenated versus standard cold perfusion preservation in kidney transplantation (COMPARE): a randomised, double-blind, paired, phase 3 trial. Lancet. 2020 Nov 21;396(10263):1653-1662. doi: 10.1016/S0140-6736(20)32411-9. PMID 33220737
- [Background] Sarkar M, Prabhu V. Basics of cardiopulmonary bypass. Indian J Anaesth. 2017 Sep;61(9):760-767. doi: 10.4103/ija.IJA_379_17. PMID 28970635
- [Background] Wang X, Zhang J, Feng K, Yang Y, Qi W, Martinez-Vazquez P, Zhao G, Wang T. The effect of hypothermia during cardiopulmonary bypass on three electro-encephalographic indices assessing analgesia and hypnosis during anesthesia: consciousness index, nociception index, and bispectral index. Perfusion. 2020 Mar;35(2):154-162. doi: 10.1177/0267659119864821. Epub 2019 Aug 7. PMID 31387454